CLINICAL TRIAL: NCT06255093
Title: You & Me Healthy: Youth Empowered Self-Care Substudy (YES)
Acronym: YES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Miami-Dade County Parks and Recreation (Other); Durham Parks and Recreation (Durham, NC) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00114773
Record Dates: First submitted 2024-02-05; First posted 2024-02-12 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-06

CONDITIONS: Anxiety; Wellness, Psychological
Keywords: Anxiety; Mental Health; Psychological Wellness; Recreational Activities; Community programs; School-aged Youth; Parks and Recreation; Afterschool Activities
MeSH Terms: conditions — Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants will be self-triaged to one of two study arms: (1) Pre-surveys only (did not meet referral criteria based on screening assessment) and receive online mental wellness education and anxiety treatment options information; (2) Pre-surveys, meet referral criteria, referred to a program, post-surveys. Post-surveys will occur at the end of the out-of-school program, or 4 months after joining the program (whichever comes first).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Surveys Only (Other): Pre-surveys only (did not meet referral criteria based on screening assessment) and receive online wellness education and anxiety treatment options information
  Interventions: Behavioral: Pre-surveys only
- Pre-Surveys, Recreational Program Referral, Post Surveys (Other): Pre-surveys, meet referral criteria, referred to a program, post-surveys. Post-surveys will occur at the end of the out-of-school program, or 4 months after joining the program (whichever comes first).
  Interventions: Behavioral: Community-based recreation program referral

INTERVENTIONS:
Behavioral: Community-based recreation program referral — Provide referral to local Parks and Recreation for programs of interest and participation. Participants will have the option to join a program (up to 4months) and have access to additional resources via study webpage to identify support services.
  Arms: Pre-Surveys, Recreational Program Referral, Post Surveys
Behavioral: Pre-surveys only — Receive online wellness education and anxiety treatment options information
  Arms: Pre-Surveys Only

SUMMARY:
You & Me Healthy: Youth Empowered Self-Care, or YES, is a study that aims to link 150 youth ages 8-12 and families to free or low-cost community-based programs, resources, and clinical care options that promote mental wellness and help reduce anxiety.

Community-based programs can include:

* Afterschool programs
* Local parks and recreation activities
* Youth social programming

DETAILED DESCRIPTION:
The You & Me Healthy; Youth Empowered Self-care study seeks to evaluate a direct-to-participant mental health intervention for youth living in underserved communities, comprising online self-screening tools, educational materials and online linkage to treatment options, and referral to free or low-cost accessible out-of-school community-based resources. Participants will self-'triage' online to access education, community resources, and clinical care options when necessary. This work will provide access and explore mechanisms for addressing wellness and anxiety needs among youth drawing from self-reported and web interaction data over a 4-month period. The central hypothesis is that the researchers will demonstrate the value of a direct-to-participant, community asset based mental health promotion program in response to COVID-19 impacts. In addition, the team aims to specifically identify approaches to enable access to community-based anxiety and mental wellness resources in underserved populations.

Out-of-school youth programs play an important role in supporting students' mental health, yet program participation has dwindled since the COVID-19 pandemic. These programs provide students with psychosocial, developmental, and health and wellness benefits. Specifically, structured youth programs can engage students in recreation, provide academic enrichment, access to green spaces, as well as opportunities for promoting social interaction and connectedness with peers, adaptive functioning, mentorship, as well as resilience, mental health, and well-being. Out-of-school youth programs are particularly critical for students who live in under resourced communities with high transportation vulnerability and limited access to community-based recreation, although unmet demand for programs is highest in underserved areas. Nationally, 9 out of 10 parents agree that out-of-school youth programs are important to their community, and 80% of North Carolina parents indicate that these programs give them peace of mind and help them to keep their jobs. Out-of-school youth programs also have been proposed as an ideal setting for supporting children's health and wellness. Put simply, out-of-school youth programs provide students with safe and supportive settings for recreation, mentorship, learning, and structure that are particularly essential for underserved communities. However, the COVID-19 pandemic has created hardships for youth to attend out-of-school programs nationwide. Prior to the COVID-19 pandemic, over 10 million youth participated in out-of-school programs nationally, although more than 80% of programs reported difficulties providing ongoing services during the COVID-19 pandemic due to poor enrollment. The gap in psychosocial support typically provided through out-of-school youth programs has likely exacerbated mental health needs during the pandemic, particularly for underserved students, and further overburdening the health care system.

The research team is working together with two large community organizations as partners for this study (Durham Parks and Recreation Department and Miami-Dade County Parks and Recreation Department), who will coordinate directly with 150 youth and families (75 participants per site) to link youth to community-based youth programs that have potential to support youth mental health needs. All eligible and consented participants will complete basic data collection including demographics, mental health symptom questions, additional barriers to program enrollment and attendance, and satisfaction survey questions using REDCap. Participants will also receive online resource linkage to mental wellness education and anxiety treatment locations as applicable.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, an individual must meet all of the following criteria:

  1. Self-reported primary residence within the pre-identified communities
  2. Age 8-12 years at enrollment
  3. Provision of signed and dated informed consent form

Exclusion Criteria:

* There are no exclusion criteria for this study if all above inclusion criteria are met.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants referred to youth community-based programs with potential to promote mental health that are free/low-cost | Up to 4 months
Number of youth community-based programs with potential to promote mental wellness offered that are free/low-cost (self-reported) | Up to 4 months
Number of youth enrollees to community-based programs with potential to promote mental wellness that are free/low-cost (self-reported) | Up to 4 months
Number of consented participants who complete self-screening assessment | Baseline
Proportion of consented participants who complete self-screening assessment | Baseline
Proportion of participants who visited the online resources page | Up to 4 months
Change in anxiety symptoms, as measured by survey | Baseline, up to 6 months
  Scale: Screen for Child Anxiety Related Emotional Disorders (SCARED) Survey- Parent Version
Change in mental wellness needs, as measured by survey | Baseline, up to 6 months
  KIDSCREEN #27- Health Screen QUestionnaire for Children and Young People ( Parent version)

OTHER OUTCOMES:
Barriers to youth program enrollment and attendance, as measured by post-participation survey | Up to 6 months
Participant Satisfaction, as measured by participant satisfaction survey | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Emily D'agostino, DPH, Principal Investigator — Duke University; Christoph Horniik, MD, PhD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Miami-Dade County Parks and Recreation, Miami, Florida
  - Durham Parks and Recreation, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] D'Agostino EM, Frazier SL, Hansen E, Patel HH, Ahmed Z, Okeke D, Nardi MI, Messiah SE. Two-Year Changes in Neighborhood Juvenile Arrests After Implementation of a Park-Based Afterschool Mental Health Promotion Program in Miami-Dade County, Florida, 2015-2017. Am J Public Health. 2019 Jun;109(S3):S214-S220. doi: 10.2105/AJPH.2019.305050. PMID 31241997
- [Background] Frazier SL, Cappella E, Atkins MS. Linking mental health and after school systems for children in urban poverty: preventing problems, promoting possibilities. Adm Policy Ment Health. 2007 Jul;34(4):389-99. doi: 10.1007/s10488-007-0118-y. Epub 2007 Mar 6. PMID 17340183
- [Background] Frazier SL, Dinizulu SM, Rusch D, Boustani MM, Mehta TG, Reitz K. Building Resilience After School for Early Adolescents in Urban Poverty: Open Trial of Leaders @ Play. Adm Policy Ment Health. 2015 Nov;42(6):723-36. doi: 10.1007/s10488-014-0608-7. PMID 25425012
- [Background] Frazier SL, Mehta TG, Atkins MS, Hur K, Rusch D. Not just a walk in the park: efficacy to effectiveness for after school programs in communities of concentrated urban poverty. Adm Policy Ment Health. 2013 Sep;40(5):406-18. doi: 10.1007/s10488-012-0432-x. PMID 22843303
- [Background] Frazier SL, Rusch D, Coxe S, Stout TJ, Helseth SA, Dirks MA, Bustamante EE, Atkins MS, Glisson C, Green PD, Bhaumik D, Bhaumik R. After-School Programs and Children's Mental Health: Organizational Social Context, Program Quality, and Children's Social Behavior. J Clin Child Adolesc Psychol. 2021 Mar-Apr;50(2):215-228. doi: 10.1080/15374416.2019.1683849. Epub 2020 Feb 14. PMID 32058822
- [Background] Goodman AC, Ouellette RR, D'Agostino EM, Hansen E, Lee T, Frazier SL. Promoting healthy trajectories for urban middle school youth through county-funded, parks-based after-school programming. J Community Psychol. 2021 Sep;49(7):2795-2817. doi: 10.1002/jcop.22587. Epub 2021 Apr 29. PMID 33914915
- [Background] Hedemann ER, Frazier SL. Leveraging After-School Programs to Minimize Risks for Internalizing Symptoms Among Urban Youth: Weaving Together Music Education and Social Development. Adm Policy Ment Health. 2017 Sep;44(5):756-770. doi: 10.1007/s10488-016-0758-x. PMID 27544670
- [Background] Jennings V, Baptiste AK, Osborne Jelks N, Skeete R. Urban Green Space and the Pursuit of Health Equity in Parts of the United States. Int J Environ Res Public Health. 2017 Nov 22;14(11):1432. doi: 10.3390/ijerph14111432. PMID 29165367
- [Background] Jones SE, Ethier KA, Hertz M, DeGue S, Le VD, Thornton J, Lim C, Dittus PJ, Geda S. Mental Health, Suicidality, and Connectedness Among High School Students During the COVID-19 Pandemic - Adolescent Behaviors and Experiences Survey, United States, January-June 2021. MMWR Suppl. 2022 Apr 1;71(3):16-21. doi: 10.15585/mmwr.su7103a3. PMID 35358165
- [Background] McCormick R. Does Access to Green Space Impact the Mental Well-being of Children: A Systematic Review. J Pediatr Nurs. 2017 Nov-Dec;37:3-7. doi: 10.1016/j.pedn.2017.08.027. Epub 2017 Sep 4. PMID 28882650
- [Background] Parenteau AM, Boyer CJ, Campos LJ, Carranza AF, Deer LK, Hartman DT, Bidwell JT, Hostinar CE. A review of mental health disparities during COVID-19: Evidence, mechanisms, and policy recommendations for promoting societal resilience. Dev Psychopathol. 2023 Oct;35(4):1821-1842. doi: 10.1017/S0954579422000499. Epub 2022 Sep 13. PMID 36097815
- [Background] Racine N, McArthur BA, Cooke JE, Eirich R, Zhu J, Madigan S. Global Prevalence of Depressive and Anxiety Symptoms in Children and Adolescents During COVID-19: A Meta-analysis. JAMA Pediatr. 2021 Nov 1;175(11):1142-1150. doi: 10.1001/jamapediatrics.2021.2482. PMID 34369987
- [Background] Saltzman LY, Lesen AE, Henry V, Hansel TC, Bordnick PS. COVID-19 Mental Health Disparities. Health Secur. 2021 Jun;19(S1):S5-S13. doi: 10.1089/hs.2021.0017. Epub 2021 May 19. PMID 34014118
- [Background] Twohig-Bennett C, Jones A. The health benefits of the great outdoors: A systematic review and meta-analysis of greenspace exposure and health outcomes. Environ Res. 2018 Oct;166:628-637. doi: 10.1016/j.envres.2018.06.030. Epub 2018 Jul 5. PMID 29982151
- See also: Afterschool in the time of COVID-19. — http://afterschoolalliance.org/documents/Afterschool-COVID-19-Wave-1-Fact-Sheet.pdf
- See also: Centers for Disease Control and Prevention. (2023). COVID-19 Provisional Counts - Health Disparities — http://www.cdc.gov/nchs/nvss/vsrr/covid19/health_disparities.htm
- See also: Inspiring Learning. Safe and Supportive. Lifeline for Working Families. This is Afterschool in North Carolina — http://www.afterschoolalliance.org/documents/nc-afterschool-facts.pdf
- See also: New Household Survey: North Carolina Is a 'Top 10 State for Afterschool, ' Even as Unmet Demand for Programs Increases — http://www.ncforum.org/new-household-survey-north-carolina-is-a-top-10-state-for-afterschool-even-as-unmet-demand-for-programs-increases/
- See also: United States of America: Who coronavirus disease (covid-19) dashboard with vaccination data. — http://covid19.who.int/region/amro/country/us